CLINICAL TRIAL: NCT06529367
Title: Comparing a Home Vision Self-Assessment Test to Office-Based Snellen Visual Acuity in Myopic Children
Status: Recruiting | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ahmed Ali Amer, Lecturer of Ophthalmology, Faculty of Medicine, South Valley University, Qena, Egypt., South Valley University
Other Study IDs: SVU\MED\OPH026/4/24/7/887
Record Dates: First submitted 2024-07-27; First posted 2024-07-31 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Home Vision; Office-Based Snellen Visual Acuity; Myopic Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Visual Acuity Testing group: Home vision assessment will be conducted using the "Letter Distance Chart" PDF document, a modified Early Treatment of Diabetic Retinopathy Study (ETDRS) chart for testing at 5 or 10 feet, and released for public use.
  Patients will be asked to use the 5-foot distance for standardization, which allows for visual acuity assessment from 20/16 to 20/200.
  Patients will be asked to wear their current corrective lens for distance, to take the test at home in a place with good lighting, and to test each eye separately.
  Office-based vision testing will be performed by a trained ophthalmic technician in a dimmed room with the Snellen chart illuminated on a screen. Patients will be asked to wear their current corrective lens for distance and an eye occluder will be used to test each eye separately.
  Interventions: Other: Snellen chart

INTERVENTIONS:
Other: Snellen chart — Patients will be asked to use the 5 feet distance for standardization, which allows for visual acuity assessment from 20/16 to 20/200.
  Patients will be asked to wear their current corrective lens for distance, to take the test at home in a place with good lighting and to test each eye separately.
  Office-based vision testing will be performed by a trained ophthalmic technician in a dimmed room with the Snellen chart illuminated on a screen. Patients will be asked to wear their current corrective lens for distance and an eye occluder will be used to test each eye separately.

SUMMARY:
This study aims to compare a home vision self-assessment test to office-based Snellen visual acuity in myopic children.

DETAILED DESCRIPTION:
Visual impairment is an important public health issue worldwide, with a heavy socioeconomic burden. More than 400 million people globally have mild to severe visual impairment.

Visual acuity (VA) screening is the most basic part of ophthalmic examination. Home vision screening tests have become an important way to obtain a measure of an individual's VA without an office-based clinic visit. Knowing a patient's VA can help ophthalmologists remotely triage acute calls, monitor visual recovery after medical or surgical interventions, and ensure visual stability in follow-up telemedicine visits.

Home vision screening tests have become an important way to obtain a measure of an individual's VA without an office-based clinic visit. Numerous electronic home vision assessment tools exist, but many of these are used through applications on mobile or tablet devices.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 18 years.
* Both sexes.
* Patients who completed the home visual acuity test and have a subsequent office-based visual acuity test.

Exclusion Criteria:

* Last in-office visual acuity of 20/125 or worse in both eyes (to allow for a buffer of at least 2 lines of vision from the upper limit of 20/200 on the home vision assessment).
* Lack of access to MyChart.
* History of keratopathy, cataract, glaucoma, retinal detachment, neuro-ophthalmic disease, or other eye diseases.
* History of ophthalmic surgery or trauma.
* History of systemic diseases.
* Severe psychological or psychiatric diseases.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This cross-sectional study will be carried out on 80 myopic children aged ≤ 18 years, who completed the home visual acuity test and have a subsequent office-based VA test at South Valley University for a period from July 2024 to January 2025 after approval from the institutional ethical committee.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Agreement of visual acuity between office and home | immediately after test performing
  Agreement of visual acuity between office and home will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley University, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.